CLINICAL TRIAL: NCT01518933
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of LEGALON SIL for the Treatment of HCV Recurrence in Stable Liver Transplanted Patients
Brief Title: Effect of LEGALON SIL on Hepatitis C Virus Recurrence in Stable Liver Transplanted Patients
Acronym: LEG-SIL-LTX-02
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: when a blind review highlighted that at least 43% of patients had a virological response
Sponsor: Rottapharm (Industry)
Collaborators: Azienda Ospedaliera Universitaria Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEG-SIL-LTX-02
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis C Virus Recurrence
Keywords: HCV recurrence; stable liver transplanted patients
MeSH Terms: interventions — Silybin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silibilin (Legalon-SIL) (Experimental): 20 mg/kg Silibinin (Legalon SIL) ,as per randomization schedule, will be administered daily as a 2-h infusion for 14 days.
  Interventions: Drug: Silibinin (Legalon-SIL)
- Saline (Placebo Comparator): Placebo (saline), as per randomization schedule, will be administered daily as a 2-h infusion for 14 days.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Silibinin (Legalon-SIL) — 20 mg/kg Silibinin (Legalon SIL), as per randomization schedule, will be administered daily as a 2-h infusion for 14 days.
  Other Names: Legalon-SIL; SHS
  Arms: Silibilin (Legalon-SIL)
Drug: Saline — Placebo
  Other Names: Placebo (saline), as per randomization schedule, will be administered daily as a 2-h infusion for 14 days
  Arms: Saline

SUMMARY:
Hepatitis C virus (HCV)-related liver disease is the most common indication for liver transplantation (LT). However, LT does not cure the infection, and therapeutic strategies resulted in very limited efficacy and tolerability in LT recipients. In view of its postulated safety profile, Silibinin seems an ideal drug to be used in the setting of HCV recurrent patients after liver transplantation.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV)-related liver disease continues to be the most common indication for liver transplantation (LT) in both the United States and Europe. However, LT does not cure the infection, and re-infection of the liver allograft universally occurs. Recurrent HCV hepatitis often follows an accelerated course after LT, and histological recurrence occurs in approximately 50% of patients within 1 year after LT; 15-30% of them develop cirrhosis within 5 years. In this context, a peculiar feature is represented by the rapid course of liver fibrosis. Therapeutic strategies for managing the primary cause of liver damage, i.e. HCV infection, irrespective of application in pre-, peri-, and/or post-LT periods resulted in very limited efficacy and tolerability in LT recipients.

In view of its postulated safety profile, Silibinin seems an ideal drug to be used in the setting of HCV recurrent patients after liver transplantation.

Silibinin, a flavonolignan representing the main component (60%) of Silymarin and proposed as an anti-hepatotoxic agent for the treatment of various liver diseases has been recently reported to beneficially modulate the pro-fibrogenic potential of HSC, thus representing a very attractive possibility in the transplanted population. Besides the anti-inflammatory properties, Silibinin is able to inhibit Tumor necrosis factor-alpha (TNF-α). This is a proinflammatory cytokine with a major role in both acute and chronic viral, bacterial and fungal infections.

The primary objective is to determine the effect of post-transplant treatment with Legalon SIL on HCV viral load 30 days after the beginning of treatment.

44 stable liver transplanted patients with HCV recurrence will be randomized 3:1 to receive Legalon-SIL or Placebo. Randomized patients will be treated for 14 consecutive days with Legalon-SIL or Placebo. Patients dropping-out before the end of treatment period will be replaced.

Patients will be followed up for 1 year to monitor the effect of treatment on liver fibrosis, liver functional state, lymphocyte activation, and viral load.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide signed and dated informed consent before undergoing any trial related procedure.
* Males or females aged ≥ 18 and ≤ 70.
* Patients with HCV recurrent chronic hepatitis after liver transplantation, not responding to treatment with peginterferon/ribavirin (i.e. the so called standard of care, SOC).
* Stable (≥ 1 year) liver transplanted patients with HCV recurrence (as indicated by positive serum HCV-RNA, increase in transaminases, signs of graft damage according to HCV recurrence and/or presence of liver fibrosis as assessed by Fibroscan).
* Patients without biochemical, clinical and/or histological suspicion of rejection.
* Patients must be able to communicate, participate and comply with the requirements of the entire study.
* Female patients of child-bearing potential must agree on using a contraceptive method (oral contraceptive, intra-uterine device [IUD], transdermal contraceptive patch) and must have a negative pregnancy test at screening.

Exclusion Criteria:

* Patients with active hepatocellular carcinoma or other neoplasia (excluding cutaneous carcinoma in view of the high prevalence in the transplanted population).
* Patients with active biliary tract anomalies.
* Patients with a rejection episode in the 6 months preceding study inclusion.
* Patients on active interferon treatment.
* Female patients who are pregnant or breast-feeding.
* Patients with clinically significant laboratory abnormalities at screening.
* Patients with creatinine clearance < 50 ml.
* Patients with any abnormality on physical examination, vital signs (sitting systolic blood pressure greater than 140 mmHg, sitting diastolic blood pressure greater than 90 mmHg and pulse greater than 80 bpm) and ECG, unless these abnormalities are judged to be not clinically significant by the Investigator (a note about this must be made on the electronic Case Report Form - e-CRF).
* Patients taking any concomitant medication that is not allowed and that cannot be discontinued for the entire study period.
* Patients who are already taking other investigational drugs/treatments or have taken part in a clinical study within the previous 3 months or 5 half lives (whichever is longer).
* Patients with known hypersensitivity to any of the test materials or related compounds.
* Patients with a history of drug, alcohol or other substance abuse or other factors limiting their ability to co-operate during the study.
* Patients not available to attend all the test days and investigations as foreseen by the protocol, or unable to understand the aim, procedure or possible hazards of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Viral load | 30 days after the beginning of treatment
  To determine the effect of post-transplant treatment with Legalon SIL on HCV viral load 30 days after the beginning of treatment.

SECONDARY OUTCOMES:
Viral load and lymphocyte activation | 1 year after the beginning of the treatment
  To determine the effect of post-transplant treatment with Legalon SIL on HCV viral load and lymphocyte activation one year after the beginning of treatment.
Fibrosis | 1 year after the beginning of the treatment
  To determine the effect of post-transplant treatment with Legalon SIL on fibrosis and functional state.
Safety | 1 year
  To determine the safety and tolerability of post-transplant treatment with Legalon SIL, including evaluation of its effect on the levels of immunomodulators.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Di Leo, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Policlinico Consorziale - Bari
Locations (1):
- Azienda Ospedaliero-Universitaria Policlinico Consorziale, Bari, Bari, Italy

REFERENCES:
- [Derived] Rendina M, D'Amato M, Castellaneta A, Castellaneta NM, Brambilla N, Giacovelli G, Rovati L, Rizzi SF, Zappimbulso M, Bringiotti RS, Di Leo A. Antiviral activity and safety profile of silibinin in HCV patients with advanced fibrosis after liver transplantation: a randomized clinical trial. Transpl Int. 2014 Jul;27(7):696-704. doi: 10.1111/tri.12324. Epub 2014 May 10. PMID 24673819